CLINICAL TRIAL: NCT07187219
Title: Efficacy of Repetitive Transcranial Magnetic Stimulation Over the Primary Cortex in Patients With Neuropathic Pain and Cancer: Cross-over and Placebo-control Study
Brief Title: Efficacy of Repetitive Transcranial Magnetic Stimulation Over the Primary Cortex in Patients With Neuropathic Pain and Cancer
Acronym: NeuroCanPain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24CH024; 2024-A01195-42 (Other: ANSM)
Record Dates: First submitted 2025-06-18; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Chronic Neuropathic Pain
Keywords: Neuropathic pain; Cancer; Transcranial magnetic stimulation; Neuromodulation; Pain relief
MeSH Terms: conditions — Neoplasms; Neuralgia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This project is a cross-over, double-blinded, and placebo-control study, including 5 sessions of either M1 or "sham" rTMS, a wash-out period (8 weeks), followed by 5 sessions of the other stimulation option (I.e., two arms: M1-sham or sham-M1; order randomized between patients).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active rTMS - Sham (Experimental): 5 stimulation sessions on M1 - washout 8 weeks - 5 sham stimulation sessions (placebo-control, same site, inactive stimulation)
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS) - active; Device: Repetitive transcranial magnetic stimulation (rTMS) - inactive
- Sham - Active rTMS (Experimental): 5 sham stimulation sessions (placebo-control, same site, inactive stimulation) - washout 8 weeks - 5 stimulation sessions on M1
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS) - active; Device: Repetitive transcranial magnetic stimulation (rTMS) - inactive

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation (rTMS) - active — rTMS session active on the primary motor cortex
Device: Repetitive transcranial magnetic stimulation (rTMS) - inactive — rTMS session inactive on the primary motor cortex

SUMMARY:
High-frequency repetitive transcranial magnetic stimulation (rTMS) of the primary motor cortex (M1) has shown its efficacy to alleviate pain in patients suffering from refractory neuropathic pain. rTMS is now considered as 3rd-line therapy (by the French Society for the Study and Treatment of Pain) for patient's refractory to drug therapy.

However, its efficacy in chronic neuropathic pain related to cancer has not yet been specifically studied, and it therefore remains relatively inaccessible for these patients. This project is a cross-over, double-blinded, and placebo-control study, including 5 sessions of either M1 or "sham" rTMS, a wash-out period (8 weeks), followed by 5 sessions of the other stimulation option (I.e., two arms: M1-sham or sham-M1; order randomized between patients). Treatment efficacy will be assessed in comparison to the placebo condition. Primary outcome is the percentage of pain relief between active and sham rTMS. Other variables to describe quality of life, sensory, neuropathic, and mood states as well as resting-state fMRI will be collected before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated to or entitled under a social security scheme
* Patient who has received informed information about the study and who has co-signed, with the investigator, a consent form to participate in the study.
* Patient aged 18 to 85 (male or female),
* Central or peripheral neuropathic pain related to cancer and/or its treatment;
* Chronic pain (present for more than 4 months) whose intensity is greater than or equal to 4/10 on a VAS (Visual Analogue Scale) numerical scale.
* Pain present on a daily or almost daily basis (at least 4 days a week)
* Patient not completely relieved by recommended first- and second-line drug treatments for neuropathic pain
* Stable analgesic treatment (no new treatment or dosage adjustment) for at least one month and will not need to be modified for the duration of the study.
* Patient can be followed throughout the study.
* Indication for rTMS of the motor cortex by a neurologist.

Exclusion Criteria:

* Accident at work or litigation,
* Contraindication to rTMS or MRI (treatment with seismotherapy during the previous month; history of cranial trauma; intracranial hypertension; intracerebral metal clip; piercing; pacemaker; insulin pump; metal prosthesis; pregnant or breast-feeding woman; claustrophobia).
* Chronic alcoholism
* Abuse of drugs or psychoactive substances
* Neuropathic pain as part of a progressive pathology (e.g. HIV),
* Presence of other pain of greater intensity than the neuropathic pain leading to inclusion
* Acute stroke (< 3 months)
* Patient with brain tumour lesions
* Patient with infectious or metabolic brain lesions
* Patients with severe or recent cardiac disorders
* Patients with cognitive impairment
* Patient unable to understand informed consent,
* Patients refusing to stop or unable to stop treatments prohibited during the study, such as morphine.
* Patients participating in another research protocol involving a medicinal product within 30 days prior to inclusion.
* Patients deprived of their liberty or under legal protection (guardianship, curatorship, safeguard of justice, family habilitation).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
PAIN RELIEF | Week 7 after the start of RTMs stimulation
  PAIN from 0% : no pain relief at all to 100%: completely relief.

SECONDARY OUTCOMES:
Pain Intensity with Visual analog scale (VAS) | day 7 post RTMs stimulation
  0 no pain to 10 extremely pain
score of Neuropathic Pain Symptom Inventory - NPSI | day 7 post RTMs stimulation
  [0= zero neuropatthic pain to 100= maximum neuropathic pain]
Brief Pain Inventory - BPI | day 7 post RTMs stimulation
  1 - 4 = Mild Pain. 5 =Worst Pain Score 6 = Moderate Pain. 7=Worst Pain Score 10 = Severe Pain.
Pain relief | day 7 post RTMs stimulation
  scale ranging from 0% = no relief to 100% = fully relieved
Visual Analogic Scale VAS on emotional dimension of pain | day 7 post RTMs stimulation
  Visual Analogic Scale VAS (0 = not unpleasant) to 10 = extremely unpleasant)
Visual Analogic Scale (VAS) on attentional dimension of pain | day 7 post RTMs stimulation
  0 = does not attract at all to 10 = completely attracts
consumption of rescue analgesics | Week 7 after the start of RTMs stimlulation
Effect of rTMS on quality of life | Week 7 after the start of RTMs stimlulation
  Quality of life score (EQ-5D) from 0 to 100. 100 corresponds to the best health.
HADS: Hospital Anxiety and Depression Scale | Week 7 after the start of RTMs stimlulation
  from 0 to 14: no anxiety disorders; from 15 to 42: existence of anxiety disorders.
Tolerance | week 7 after the start of RTMs stimulation
  Tolerance will be defined as the absence of adverse effects throughout the duration of the protocol, as reported in systematic questionnaires."

CONTACTS AND LOCATIONS:
Overall Officials: Roland PEYRON, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- PEYRON Roland, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No